CLINICAL TRIAL: NCT04009772
Title: Single Dose Cefepime Versus Cefuroxime Plus Metronidazole as a Prophylactic Antibiotic: A Randomized Controlled Study
Brief Title: Single Dose Cefepime Versus Cefuroxime Plus Metronidazole as a Prophylactic Antibiotic During Emergency Intrapartum Cesarean Section
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Collaborators: Yasser Esmat Mohammed (Unknown)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Consultant of Obstetrics and gynecology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Antibiotic CS
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Emergency Cesarean Section; Infection Wound
Keywords: Cefepime, Cefuroxime, Metronidazole, Cesarean, Intrapartum
MeSH Terms: conditions — Wound Infection | interventions — Cefepime; Cefuroxime; Metronidazole; cefuroxime axetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Cefepime" , "Maxipime®" 1 gm (Active Comparator): Patient will receive "Cefepime" ,"Maxipime®" 1 gm IV during cesarean section just before skin incision
  Interventions: Drug: Cefepime
- "Cefuroxime", "Zinnat®" 1gm plus "metronidazole"Flagyl®" 500 (Active Comparator): Patient will receive "Cefuroxime", "Zinnat®" 1gm ,and "metronidazole"Flagyl®" 500 IV; just before skin incision for emergency cesarean section
  Interventions: Drug: Cefuroxime plus Metronidazole

INTERVENTIONS:
Drug: Cefepime — Antibiotic prophylaxis
  Other Names: Maxipime
  Arms: "Cefepime" , "Maxipime®" 1 gm
Drug: Cefuroxime plus Metronidazole — Antibiotic prophylaxis
  Other Names: Zinnat plus Flagyl
  Arms: "Cefuroxime", "Zinnat®" 1gm plus "metronidazole"Flagyl®" 500

SUMMARY:
Compare between cefepime versus routine antibiotics as a prophylactic antibiotic during emergency cesarean section in a tertiary center of obstetric care

DETAILED DESCRIPTION:
This is a randomized double blinded study which compare between single dose cefepime versus cefuroxime plus metronidazole during emergency intrapartum cesarean section.

Outcomes will include fever, wound infection, and urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* intrapartum caesarean section

Exclusion Criteria:

* evidence of infection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site wound infection | one week
  Examining the wound after one week of the surgery to detect any infection

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No